CLINICAL TRIAL: NCT04799288
Title: Phase I/II Study of Teriflunomide in HTLV-1 Associated Myelopathy/Tropical Spastic Paraparesis
Brief Title: Teriflunomide in HTLV-1 Associated Myelopathy/Tropical Spastic Paraparesis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210016; 21-N-0016
Record Dates: First submitted 2021-03-13; First posted 2021-03-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12-18

CONDITIONS: HAM/TSP
Keywords: Aubagio; Single center; Open Label
MeSH Terms: interventions — teriflunomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teriflunomide (Experimental): Teriflunomide 14 mg daily
  Interventions: Drug: Teriflunomide

INTERVENTIONS:
Drug: Teriflunomide — Teriflunomide 14mg will be administered orally as 1 tablet once daily during the 9-month treatment phase of the study.

SUMMARY:
Background:

HTLV-1 associated myelopathy/tropical spastic paraparesis (HAM/TSP) is a rare, progressive disease. It occurs in some people infected with the HTLV-1 virus. It leads to weakness in the lower limbs and other serious problems. It has no treatment. Teriflunomide is a drug used to treat multiple sclerosis. It reduces immune cells that make the disease worse. Researchers want to learn if this drug can help people with HAM/TSP.

Objective:

To learn the effects, immune response, safety, and tolerability of teriflunomide in people with HAM/TSP.

Eligibility:

Adults ages 18 and older with HAM/TSP.

Design:

Participants will be screened under protocol 98-N-0047.

Participants will have a medical history. They will have physical and neurological exams. They will have blood and urine tests.

Participants will take 1 tablet of the study drug once a day for 9 months. They will keep a drug diary.

Participants will have lymphapheresis. For this, blood is drawn from a needle in one arm. A machine divides the blood into red cells, plasma, and white cells. The white cells are removed. The plasma and red cells are returned to the participant through a needle in the other arm.

Participants will have lumbar punctures ( spinal taps ). For this, a thin needle is inserted into the spinal canal in the lower back. Spinal fluid is removed.

Participants will have magnetic resonance imaging (MRI) of the brain and spine. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the MRI, participants will lie on a table that can slide in and out of the scanner.

Participation will last for 15 months.

DETAILED DESCRIPTION:
Study Description:

In this single center, single arm, open label, baseline versus treatment pilot clinical trial, sixteen subjects with HAM/TSP will receive teriflunomide 14mg by mouth once a day in an initial 9 month treatment phase, followed by a 3 month post treatment follow-up phase. Outcome measures will be collected every 3 months for the duration of the study.

Objectives:

We will determine the effects of teriflunomide, an FDA approved drug for the treatment of relapsing remitting multiple sclerosis that inhibits de novo pyrimidine synthesis, on immune activation markers in patients with HAM/TSP and the correlation of these with virological, radiological and clinical measures of disease burden .

Endpoints:

The primary outcome measure is ex vivo spontaneous lymphoproliferation in HAM/TSP patients receiving teriflunomide. Secondary outcome measures will include determination of immune activation patterns of PBMC and CSF using multicolor flow cytometric analysis and HTLV-I proviral load in blood and CSF. Safety and tolerability of teriflunomide will be assessed by tabulation of adverse events, clinical exam, standardized neurological disability scales (EDSS, IPEC, HAQ-DI), MR imaging of brain and spinal cord and clinical laboratory studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* 18 years or older
* Diagnosis of HAM/TSP as defined by WHO criteria, including a positive HTLV-1 EIA and confirmatory Western Blot.
* Enrolled in 98-N-0047
* Patient must be willing and able to comply with all the aspects of trial design and follow-up.
* Negative QuantiFERON-TB gold, or completion of latent tuberculosis infection treatment, per CDC and National TB Controllers Association recommendations in the event of a positive test result

  --In the event of an indeterminant result, the test will be repeated. Should two consecutive tests yield indeterminant results, a chest x-ray will be performed to rule out radiographic evidence of a latent TB infection. Negative imaging will enable the subject to qualify for participation in the study.
* Ability to take oral medication and be willing to adhere to the protocol regimen
* Patients must be able to provide informed consent
* If able to become pregnant or to father a child, patient must agree to commit to the use of a reliable/accepted method of birth control (i.e. hormonal contraception (birth control pills, injected hormones, vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom with spermicide) or surgical sterilization (hysterectomy, tubal ligation, or vasectomy) for the duration of the treatment arm of the study and for two years following cessation of treatment with teriflunomide.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Alternative diagnoses that can explain neurological disability
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial or interfere with participation for the full duration of the trial; or not in the best interest of the subject to participate, in the opinion of the treating investigator
* Severe immunodeficiency, bone marrow disease, or severe, uncontrolled infections.
* Liver dysfunction, as indicated by baseline aspartate aminotransferase (AST) or alanine or alanine aminotransferase (ALT) greater than 2 times the upper limit of normal
* Positive serological evidence of HIV, HTLV-II, Hepatitis B or C
* Treatment with immunomodulatory/immunosuppressive therapy is exclusionary except in the cases below:

  * current use of topical steroids
  * Study participants who have been prescribed <= 10 mg prednisone (PO) per day will be required to discontinue this medication for a period of at least 3 months (90 days) prior to enrolling in 21-N-0016. Additionally, participants who have been prescribed burst therapy with an oral steroid as an outpatient over the course of <= 10 days (e.g., Medrol Dosepak [methylprednisolone]), can enroll after discontinuing burst dose oral steroids for at least 3 months.
* Pregnant or lactating women.
* Treatment with other investigational drugs within 6 months before enrollment
* Known hypersensitivity to teriflunomide or leflunomide
* Concomitant treatment with leflunomide

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
ex vivo spontaneous lymphoproliferation in HAM/TSP patients receiving teriflunomide | Percent change between Day 0 and month 9 of spontaneous proliferation.
  ex vivo spontaneous lymphoproliferation of HAM/TSP patients receiving teriflunomide and multicolor flow cytometric analysis of immune activation markers in both PBMCs and CSF

SECONDARY OUTCOMES:
Tabulation of adverse events | at each visit
  This is a first in HAM/TSP pilot study using teriflunomide thus important to monitor for any unexpected events related to worsening of disease laboratory and clinical measures.
Percent change between CD8+ and CD4+ cells in the CSF | between month -3 and month 9
  CD8 cells are thought to be immunopathogenic and drive the immune response. In vitro studies have shown a reduction of CD8+ and CD4+ cells in the presences of teriflunomide.
HTLV-1 proviral load in the peripheral blood mononuclear cells (PBMCs) | at month 9 and compared to Day 0
  HTLV-1 proviral load is a measure of the percent of infected cells and previous data suggests a correlation with disease activity.
HTLV-1 proviral load in the CSF cells | at month 9 and compared to month -3
  HTLV-1 proviral load is a measure of the percent of infected cells and previous data suggests a correlation with disease activity.
Change in IPEC score | at month 9 and compared to Day 0
  This is a first in HAM/TSP pilot study using teriflunomide thus important to monitor for any unexpected events related to worsening of clinical measures.
Change in EDSS score | at month 9 and compared to Day 0
  This is a first in HAM/TSP pilot study using teriflunomide thus important to monitor for any unexpected events related to worsening of clinical measures.
Change in 25-foot timed walk | at month 9 and compared to Day 0
  This is a first in HAM/TSP pilot study using teriflunomide thus important to monitor for any unexpected events related to worsening of clinical measures.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Jacobson, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that results in a publication
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: IPD will be shared under tech transfer agreements.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-N-0016.html